CLINICAL TRIAL: NCT07057531
Title: A Prospective Randomized Controlled Study Evaluating Lung Injury, Long-term Clinical Outcomes, and Environmental Impact of Tubeless Versus Intubated Video-Assisted Thoracic Surgery for Lung Cancer Resection
Brief Title: Tubeless VATS for Lung Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMU-TUBELESS-VATS-2025
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-06

CONDITIONS: Lung; Lung Cancer (NSCLC); VATS
Keywords: VATS; Tubeless; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubeless group (Experimental)
  Interventions: Procedure: Tubeless thoracic surgery
- Intubation group (Other)
  Interventions: Procedure: Tubeless thoracic surgery

INTERVENTIONS:
Procedure: Tubeless thoracic surgery — Tubeless thoracic surgery is a minimally invasive procedure performed without tracheal intubation or mechanical ventilation, allowing for spontaneous breathing. Anesthesia combines conscious sedation with local nerve blocks to ensure pain relief while preserving diaphragmatic movement. The surgical approach is similar to conventional video-assisted thoracic surgery (VATS), used for procedures like lung resections and mediastinal mass excisions. Post-operative care focuses on early mobilization and quick discharge.

SUMMARY:
This prospective cohort study evaluates lung injury, long-term clinical outcomes, and environmental impacts of tubeless video-assisted thoracic surgery (VATS) compared with conventional intubated VATS for lung cancer resection. The study aims to determine whether the tubeless approach reduces anesthetic exposure, minimizes lung injury, enhances patient recovery, and decreases carbon emissions, contributing toward sustainable surgical practices.

DETAILED DESCRIPTION:
Minimally invasive thoracic surgery typically relies on general anesthesia with endotracheal intubation and mechanical ventilation, practices associated with increased anesthetic exposure, ventilator-induced lung injury, and environmental burden due to anesthetic gas emissions. To address these issues, our research group developed the tubeless VATS technique, employing spontaneous ventilation under monitored anesthesia care with supraglottic airway devices, nerve blocks, and minimal use of opioids and volatile anesthetics.

This multicenter study prospectively enrolls patients undergoing elective lung cancer resection via either tubeless or conventional intubated VATS, following a standardized protocol. The primary objectives include assessing the incidence and severity of lung injury using mechanical power metrics derived from a validated machine-learning model, quantifying anesthetic drug usage, evaluating postoperative recovery and complication rates, and analyzing long-term clinical outcomes including overall survival and quality of life measures.

Additionally, the study investigates the environmental impact of each anesthesia method by quantifying reductions in carbon emissions associated with decreased consumption of inhalational anesthetics. Findings from this research could significantly influence clinical practice guidelines by demonstrating the benefits of tubeless VATS in enhancing patient safety, improving long-term clinical outcomes, and advancing sustainable surgical practices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years scheduled for elective video-assisted thoracic surgery (VATS) for confirmed or suspected lung cancer.
2. Clinical stage suitable for surgical resection (lobectomy, segmentectomy, or wedge resection).
3. American Society of Anesthesiologists (ASA) physical status classification ≤III.
4. Ability to understand and willingness to provide written informed consent.
5. Agreement to adhere to scheduled postoperative clinical follow-up assessments, including pulmonary function tests and survival status evaluations.

Exclusion Criteria:

1. Patients requiring bilateral pulmonary procedures or planned open thoracotomy.
2. History of severe cardiopulmonary disease or unstable medical conditions that contraindicate minimally invasive thoracic surgery.
3. Emergency surgery due to acute respiratory or cardiovascular instability.
4. Inability to cooperate with the planned anesthetic and surgical protocols or postoperative follow-up procedures.
5. Pregnancy or lactation at the time of enrollment.
6. Known allergy or contraindication to anesthetic agents or materials used in the study.
7. Enrollment in another interventional clinical study within the past 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Lung Injury Assessment | Intraoperative period (from anesthesia induction to the end of surgery, approximately 1 to 3 hours)
  Comparison of intraoperative mechanical power (MP) between tubeless and intubated VATS groups, quantified by a validated machine-learning model to evaluate ventilator-induced lung injury severity. Lower mechanical power indicates reduced lung stress and potential lung injury.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China